CLINICAL TRIAL: NCT01246609
Title: The Effect of Irrigation Solution Volume on Electrolytes and Acid-Base Balance in Patients Undergoing Percutaneous Lithotripsy
Brief Title: The Effect of Irrigation Solution Volume on Electrolytes and Acid-Base Balance
Status: Terminated | Type: Observational
Why Stopped: the doctor who ran this study, left
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0322-10CTIL
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Acid Base Imbalance; Percutaneous Lithotripsy
Keywords: acid base balance; Percutaneous Lithotripsy
MeSH Terms: conditions — Acid-Base Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

There are several surgical procedures in which irrigation fluids are used to enable vision and treatment in body cavities, such as hysteroscopy, arthroscopy and cystoscopy. Several solutions are used for irrigation: normal saline, glycin, mannitol, sorbitol and others. Post-operative complications, as visual disturbances, confusion and other neurologic symptoms were attributed to irrigation fluid absorption, water intoxication and hyponatremia, and are refered to as "TURP syndrome" when appearing following transurethral prostatectomy (TURP). Historically, a reduced serum sodium concentration has been used to diagnose absorption of electrolytes-free irrigating fluid during urologic procedures. However, neurologic symptoms following transurethral prostatectomy (TURP) do not correlate with blood sodium level, moreover, Hyponatremia may not be the sole or even the primary cause of the neurological manifestations of TURP syndrome. Other techniques were suggested for evaluating the volume of irrigation solution absorption though none is used routinely in the clinical setting.

Percutaneous Lithotripsy (PCNL) is a procedure used to treat patients with nephrolithiasis. In this procedure irrigation fluid is administered into the kidney and urinary tract collecting system. The solution used is normal saline. In earlier studies there was no evidence for absorption of the irrigation fluids, though medical literature on this issue is limited. However, minute changes in electrolytes and acid-base balance may indicate the opposite is true. Indeed, the volume of irrigation and duration of the procedure may have an effect as well. According to the investigators hypothesis, the change in Ph and reduction in base content in patients undergoing PCNL may be the result of irrigation fluid absorption, since chloride from the normal saline is known to cause such effect.

Methods This is an observational prospective study of consecutive 200 adult patients undergoing elective surgery of PCNL in the investigators operating rooms.

The investigators will collect data that is taken from the patient's file and routine management of these patients: age, gender, weight, pre-operative blood tests including: electrolytes, creatinine, hematocrit, ph, bicarbonate, base, length of the procedure, volume and type of irrigation fluids used, volume and type of intravenous fluids used. Post-operative blood tests will be recorded.

The investigators will compare pre and post-operative blood tests, especially ph, bicarbonate, base content, sodium. The investigators will analyse statistically the correlation between the change of each parameter (delta X) and the volume of irrigation fluids used during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult consent patients, undergoing elective percutaneous lithotripsy.

Exclusion Criteria:

* Pregnancy
* Pre-operative acid-base imbalance
* Urgent/emergent surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational prospective study of consequtive 200 adult patients undergoing elective surgery of percoutanous lithotripsy in our operating rooms.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Actual)